CLINICAL TRIAL: NCT03066297
Title: A Prospective Study to Optimize the Extent of Pulmonary Resection According to the Decision-Making Algorithm in Patients With Clinical Stage IA Non-Small Cell Lung Cancer
Brief Title: Optimal Extent of Pulmonary Resection in Clinical Stage IA Non-Small Cell Lung Cancer
Acronym: OREX-IA
Status: Active, not recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hong Kwan Kim, MD, PhD, Department of Thoracic and Cardiovascular Surgery, Samsung Medical Center
Other Study IDs: 2016-12-116
Record Dates: First submitted 2017-02-15; First posted 2017-02-28 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Stage IA Non-small Cell Lung Cancer
Keywords: Clinical stage IA non-small cell lung cancer; Lobectomy; Segmentectomy; Wedge resection; Sublobar resection; Limited resection
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Lobectomy: Lobectomy will be chosen as the extent of pulmonary resection according to the institutional decision-making algorithm
- Segmentectomy: Segmentectomy will be chosen as the extent of pulmonary resection according to the institutional decision-making algorithm
  Interventions: Procedure: Extent of pulmonary resection
- Wide wedge resection: Wide wedge resection will be chosen as the extent of pulmonary resection according to the institutional decision-making algorithm
  Interventions: Procedure: Extent of pulmonary resection

INTERVENTIONS:
Procedure: Extent of pulmonary resection — Extent of pulmonary resection selected based on the institutional decision-making algorithm
  Groups: Segmentectomy; Wide wedge resection

SUMMARY:
The investigatros hypothesized that selection of surgical procedure according to the pre-defined institutional decision-making algorithm will not compromise the treatment outcomes including overall survival and disease-free survival in participants with clinical stage IA non-small cell lung cancer.

The purpose of this study is to determine the outcome of participants with clinical stage IA NSCLC treated by 3 types of surgical resection (wide wedge resection, segmentectomy, or lobectomy) according to the institutional decision-making algorithm

The investigators are planning to enroll 1,000 participants who meet the pre-defined eligibility criteria over 5 years.

DETAILED DESCRIPTION:
1. Background

   * The standard extent of pulmonary resection for non-small cell lung cancer (NSCLC) is still lobectomy. However, recent advances in imaging technology and staging modalities and the widespread use of computed tomography (CT) screening have greatly increased the probability of detecting small-sized tumors, especially with ground-glass opacity (GGO) feature. Adenocarcinoma with GGO feature generally has a good prognosis due to its minimally invasive nature. Many studies have shown that these pathologically less invasive subtypes are associated with better prognoses compared with other subtypes such as acinar, papillary, micropapillary, and solid predominant invasive adenocarcinoma.
   * This recent change in the disease pattern of NSCLC from locally advanced and solid tumors to early and less invasive tumors with GGO features have led to a resurgence of interest in sublobar resection. Several retrospective studies have been conducted to compare the early and late outcomes including long-term survival between patients who underwent lobectomy and those who underwent sublobar resection.
   * Multiple reports have suggested that small-sized peripheral lung adenocarcinoma can be treated by sublobar resection, yielding survival rates similar to those of lobectomy. Lobectomy is considered to be too much for these less invasive tumors and sublobar resection would be sufficient for these tumors. If sublobar resection is equivalent to lobectomy in terms of their oncologic efficacy for the surgical treatment of NSCLC, the potential benefits of sublobar resection include (1) the preservation of vital lung parenchyma and pulmonary function, which may lead to improved early morbidities and mortalities and then late quality of life and (2) a chance for a second resection with a subsequent primary NSCLC.
   * However, when considering the published evidence for sublobar resection, its interpretation needs to be cautious. Since most studies were non-randomized, there may also have been selection bias in terms of preoperative patient risk factors (intentional vs. compromised sublobar resection), tumors of various histological subtypes or different tumor size in the study arms. Therefore, the results from two randomized trials of lobectomy versus sublobar resection for small-sized lung cancer currently ongoing in Japan (Japan Clinical Oncology Group [0802]) and in the United States (Cancer and Leukemia Group B [140503]) need to be awaited.
   * Based on these clinical circumstances and the published evidence, the investigators developed the decision-making algorithm regarding the surgical treatment for clinical stage IA NSCLC.
2. Hypothesis The investigators hypothesized that selection of surgical procedure according to the pre-defined institutional decision-making algorithm will not compromise the treatment outcomes including overall survival and disease-free survival in patients with clinical stage IA non-small cell lung cancer.
3. Purpose The purpose of this study is to determine the outcome of participants with clinical stage IA NSCLC treated by 3 types of surgical resection (wide wedge resection, segmentectomy, or lobectomy) according to the institutional decision-making algorithm
4. Study plan The investigators are planning to enroll 1,000 participants who meet the pre-defined eligibility criteria over 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. The following features should be fulfilled at preoperative thin-section CT scans

   * Solitary lung nodule
   * Lesion size is 3cm or less in its maximal dimension of the entire tumor
   * The center of the tumor is located in the outer third of the lung field in either the transverse, coronal, or sagittal plane
   * Lung cancer is suspected (or NSCLC if tissue diagnosis already obtained)
2. Clinical stage T1a-bN0M0 (according to 7th AJCC staging system)
3. Absence of proximal segmental or lobar bronchial involvement.
4. NSCLC must be confirmed in intraoperative frozen section biopsies or postoperative pathologic examinations if the lesion was not histologically confirmed before operation.
5. Age ≥ 18 years and < 75 years.
6. ECOG performance status 0-1.
7. The patient should have adequate cardiopulmonary reserve to tolerate lobectomy (ppo FEV1 > 40% and ppo DLCO > 40% or VO2 max > 15ml kg-1 min-1)
8. No prior chemotherapy or thoracic radiotherapy for any malignancy.
9. No prior malignancy within 5 years from study entry (except for non-melanoma skin cancer, superficial bladder cancer, thyroid cancer or carcinoma in situ of the uterine cervix).
10. The patient agrees to participate in the study and signs the informed consent form.

Exclusion Criteria:

1. Histologic diagnosis other than NSCLC (such as small cell lung cancer, carcinoid, pulmonary lymphoma, or other benign lung disease, etc).
2. Hilar or mediastinal lymph node metastasis suspected on imaging studies (CT or PET/CT) or confirmed preoperatively by EBUS or mediastinoscopy.
3. Parietal pleura, chest wall, or mediastinal invasion is confirmed intraoperatively or postoperatively.
4. M1a disease is confirmed intraoperatively or postoperatively.
5. Bilobectomy, sleeve resection, pneumonectomy, concomitant wedge resection, or concomitant thoracic procedure (including cardiac surgery) is performed.
6. Synchronous or metachronous multiple cancers (within the past 5 years).
7. Interstitial lung disease or severe pulmonary emphysema which makes it impossible to tolerate either lobectomy or sublobar resection.
8. Active bacterial or fungal infection.
9. Uncontrolled systemic disease which makes the patient medically unfit for thoracic surgery such as unstable angina, recent myocardial infarction, congestive heart failure, or end-stage renal or liver disease.
10. Serious mental illness or psychosis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are planned to undergo surgery for clinical stage IA non-small cell lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 1018 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 5 years
  the time from the date of the operation until the first recurrence or the last follow-up.

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
  the interval between the date of the operation and the date of death from any cause or the last follow-up
Rate of loco-regional recurrence | 5 years
  Loco-regional recurrence means tumor recurrence within the ipsilateral hemithorax and mediastinum
Rate of systemic recurrence | 5 years
  Systemic recurrence means tumor recurrence outside the bilateral hemithorax or mediastinum except for lung-to-lung metastasis
Postoperative FEV1 (Forced expiratory volume in 1 second; Liter) | 6 months, 12 months, 24 months, 36 months, 48 months, 60 months after operation date
  the volume exhaled during the first second of a forced expiratory maneuver started from the level of total lung capacity. This value reflects the pulmonary function of participants
Postoperative DLco (Diffusing capacity of the lung for carbon monoxide; mL/mmHg/min) | 6 months, 12 months, 24 months, 36 months, 48 months, 60 months after operation date
  the extent to which oxygen passes from the air sacs of the lungs into the blood. This value is also related to the pulmonary function of participants
C/T ratio at thin section CT scans | within 2 months prior to operation date
  C/T ratio is the consolidation/tumor ratio, which can be measured by the maximum diameter of consolidation to the maximum tumor diameter. Pathologic invasiveness of tumors can be predicted by this value.
Postoperative pathologic subtypes | 1 month after operation date
  (according to the 2015 WHO classification of lung tumors)
Incidence of lymph node metastasis | within 1 month after operation date
  The investigators will check the incidence of lymph node metastasis from the permanent pathology report.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Kwan Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No